CLINICAL TRIAL: NCT03383718
Title: Comparison of Dobutamine Stress Echocardiography and Fractional Flow Reserve in Patients With Moderate Coronary Artery Disease: Stable and Non-culprit Lesions Investigation
Brief Title: DSE vs. FFR in SCAD and BYSTANDER Lesions
Acronym: DSE-vs-FFR
Status: Completed | Type: Observational
Sponsor: Bajcsy-Zsilinszky Hospital (Other)
Collaborators: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Peter Andrassy MD.PhD., Clinical Lead of Cardiology Department, Bajcsy-Zsilinszky Hospital
Other Study IDs: 1.0
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Heart Disease
Keywords: Coronary Artery Disease; Fractional Flow Reserve; Dobutamine Stress Echocardiography; Stable Coronary Artery Disease; Bystander Coronary Artery Disease; Non-Culprit Lesions; Acute Myocardial Infarction
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DSE+/FFR+: Patients with positive Dobutamine Stress Echocardiography and with positive Fractional Flow Reserve Revascularisation
  Interventions: Procedure: Revascularisation
- DSE+/FFR- or DSE-/FFR+ or DSE-/FFR-: Patients with positive Dobutamine Stress Echocardiography and with negative Fractional Flow Reserve
  Patients with negative Dobutamine Stress Echocardiography and with positive Fractional Flow Reserve
  Patients with negative Dobutamine Stress Echocardiography and with negative Fractional Flow Reserve
  Optimal Medical Treatment/OMT
  Interventions: Other: Optimal Medical Treatment/OMT

INTERVENTIONS:
Procedure: Revascularisation — Percutaneous coronary intervention or coronary artery bypass surgery
  Other Names: PCI or CABG
  Groups: DSE+/FFR+
Other: Optimal Medical Treatment/OMT — Standard of care in stable coronary artery disease or after acute myocardial infarction.
  Groups: DSE+/FFR- or DSE-/FFR+ or DSE-/FFR-

SUMMARY:
Enrollment:

* Patients with stable coronary artery disease (SCAD) and moderate coronary artery stenoses (30-70 %)
* Patients with acute myocardial infarction and moderate stenosis of non-culprit arteries (NCL; BYSTANDER LESION)

Aims:

* To assess the diagnostic accuracy of dobutamine stress echocardiography (DSE) and invasive fractional flow reserve (FFR) measurement
* To assess the prognostic impact of reclassification by a mismatching negative test

Hypothesis:

* DSE and FFR have similar prognostic value in both clinical settings (SCAD and NCL)
* Considering the strong negative predictive value of both DSE and FFR, one negative test is sufficiently enough to defer revascularisation, even in the case of mismatch

DETAILED DESCRIPTION:
Easy accessibility made fractional flow reserve (FFR) a widely accepted method to evaluate myocardial ischaemia in patients with moderate coronary artery stenosis, although the prognostic value for "hard" endpoints such as myocardial infarction and cardiovascular death is equivocal.

Dobutamine stress echocardiography (DSE) is a useful and safe non-invasive functional test for myocardial ichaemia evaluation. There are robust data confirming the prognostic value of DSE regarding the same "hard" endpoints.

In patients with SCAD there are clear recommendations in the recent guidelines both for DSE guided or FFR guided revascularization but the data about prognosis is limited, especially in the case of FFR guidance. The outcome is also equivocal if there is a difference between the invasive and non-invasive test result.

In patients with acute myocardial infarction, more than 50% of patients have multivessel disease. There are clear recommendations for the management of infarct related artery, however controversy still exists for the management of angiographically moderate NCLs.

In DSE vs. FFR prospective trial, the Investigators plan to perform both the DSE and FFR tests in the above mentioned clinical settings, to investigate the correlation between them. The causes of differences between them would be investigated as well as the prognostic impact of reclassification by a second test (either DSE or FFR).

If both tests are positive, revascularisation is planned to be performed (PCI Group). In cases of either double negative or mismatching tests, optimal medical therapy will be chosen (OMT Group) with clinical follow up of at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Moderate Coronary Stenosis (30-70 %)
* Stable coronary artery disease or patients with acute myocardial infarction and at least one moderate non-culprit vessel stenosis

Exclusion Criteria:

* Left Main Coronary artery stenosis
* Age>80 years
* Known non-cardiovascular disease with poor prognosis
* Patients for whom coronary angiography or stress echocardiography is contraindicated per institutional standard of care (e.g. History of severe and/or anaphylactic contrast reaction)
* Inability to provide informed consent;
* Inability to cooperate with the investigation
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, the suitable patients have at least one moderate coronary artery stenosis identified by coronary angiography.
  There will be patients with stable coronary artery disease and patients with acute myocardial infarction having at least one non-culprit vessel stenoses.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Acute Myocardial Infarction | From baseline to at least 2 years
  Detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin (cTn)] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following: Symptoms of ischaemia. New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB).
  Development of pathological Q waves in the ECG. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
  Identification of an intracoronary thrombus by angiography or autopsy
Target Vessel Revascularisation | From baseline to at least 2 years
  The Investigated Vessel need Revascularisation because of at least Canadian Cardiology Society Angina Class III
Cardiovascular Death | From baseline to at least 2 years
  Death occurs due to Cardiovascular cause

SECONDARY OUTCOMES:
Angina | From baseline to at least 2 years
  Rehospitalisation due to Angina
Heart failure | From baseline to at least 2 years
  Rehospitalisation due to Heart Failure
Non-Cardiac Death | From baseline to at least 2 years
  Death occurs due to Non-Cardiovascular cause
Non-Target Vessel Revascularisation | From baseline to at least 2 years
  The Non-Investigated Vessel need Revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Péter Andrássy, MD.PhD., Principal Investigator — Bajcsy-Zsilinszky Hospital

IPD SHARING:
Plan to Share IPD: No
Results will be shared ONLY with the patient's other physicians.

REFERENCES:
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Christou MA, Siontis GC, Katritsis DG, Ioannidis JP. Meta-analysis of fractional flow reserve versus quantitative coronary angiography and noninvasive imaging for evaluation of myocardial ischemia. Am J Cardiol. 2007 Feb 15;99(4):450-6. doi: 10.1016/j.amjcard.2006.09.092. Epub 2006 Dec 20. PMID 17293182
- [Background] Gaibazzi N, Rigo F, Lorenzoni V, Molinaro S, Bartolomucci F, Reverberi C, Marwick TH. Comparative prediction of cardiac events by wall motion, wall motion plus coronary flow reserve, or myocardial perfusion analysis: a multicenter study of contrast stress echocardiography. JACC Cardiovasc Imaging. 2013 Jan;6(1):1-12. doi: 10.1016/j.jcmg.2012.08.009. Epub 2012 Dec 5. PMID 23219414
- [Background] Pattanshetty DJ, Bhat PK, Gandhi S, Pillai DP, Aneja A. Comparing stress testing and fractional flow reserve to evaluate presence, location and extent of ischemia in coronary artery disease. Indian Heart J. 2015 Jan-Feb;67(1):50-5. doi: 10.1016/j.ihj.2015.02.010. Epub 2015 Feb 25. PMID 25820051
- [Background] Cortigiani L, Rigo F, Gherardi S, Bovenzi F, Molinaro S, Picano E, Sicari R. Coronary flow reserve during dipyridamole stress echocardiography predicts mortality. JACC Cardiovasc Imaging. 2012 Nov;5(11):1079-85. doi: 10.1016/j.jcmg.2012.08.007. PMID 23153906
- [Background] Ojaghi-Haghighi Z, Abtahi F, Fazlolah S, Moladoust H, Maleki M, Gholami S. Coronary flow reserve, strain and strain rate imaging during pharmacological stress before and after percutaneous coronary intervention: comparison and correlation. Echocardiography. 2011 May;28(5):570-4. doi: 10.1111/j.1540-8175.2011.01366.x. Epub 2011 May 4. PMID 21539600
- [Background] Dagdelen S, Yuce M, Emiroglu Y, Ergelen M, Pala S, Tanalp AC, Izgi A, Kirma C. Correlation between the tissue Doppler, strain rate, strain imaging during the dobutamine infusion and coronary fractional flow reserve during catheterization: a comparative study. Int J Cardiol. 2005 Jun 22;102(1):127-36. doi: 10.1016/j.ijcard.2004.05.012. PMID 15939109
- [Background] Neglia D, Rovai D, Caselli C, Pietila M, Teresinska A, Aguade-Bruix S, Pizzi MN, Todiere G, Gimelli A, Schroeder S, Drosch T, Poddighe R, Casolo G, Anagnostopoulos C, Pugliese F, Rouzet F, Le Guludec D, Cappelli F, Valente S, Gensini GF, Zawaideh C, Capitanio S, Sambuceti G, Marsico F, Perrone Filardi P, Fernandez-Golfin C, Rincon LM, Graner FP, de Graaf MA, Fiechter M, Stehli J, Gaemperli O, Reyes E, Nkomo S, Maki M, Lorenzoni V, Turchetti G, Carpeggiani C, Marinelli M, Puzzuoli S, Mangione M, Marcheschi P, Mariani F, Giannessi D, Nekolla S, Lombardi M, Sicari R, Scholte AJ, Zamorano JL, Kaufmann PA, Underwood SR, Knuuti J; EVINCI Study Investigators. Detection of significant coronary artery disease by noninvasive anatomical and functional imaging. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002179. doi: 10.1161/CIRCIMAGING.114.002179. PMID 25711274
- [Background] Takx RA, Blomberg BA, El Aidi H, Habets J, de Jong PA, Nagel E, Hoffmann U, Leiner T. Diagnostic accuracy of stress myocardial perfusion imaging compared to invasive coronary angiography with fractional flow reserve meta-analysis. Circ Cardiovasc Imaging. 2015 Jan;8(1):e002666. doi: 10.1161/CIRCIMAGING.114.002666. PMID 25596143
- [Background] van der Sijde JN, Boiten HJ, van Domburg RT, Schinkel AF. Long-Term (>10 Years) Prognostic Value of Dobutamine Stress Echocardiography in a High-Risk Cohort. Am J Cardiol. 2016 Apr 1;117(7):1078-83. doi: 10.1016/j.amjcard.2016.01.002. Epub 2016 Jan 14. PMID 26839054
- [Background] Harb SC, Marwick TH. Prognostic value of stress imaging after revascularization: a systematic review of stress echocardiography and stress nuclear imaging. Am Heart J. 2014 Jan;167(1):77-85. doi: 10.1016/j.ahj.2013.07.035. Epub 2013 Nov 21. PMID 24332145
- [Background] Cortigiani L, Bigi R, Sicari R, Landi P, Bovenzi F, Picano E. Prognostic value of pharmacological stress echocardiography in diabetic and nondiabetic patients with known or suspected coronary artery disease. J Am Coll Cardiol. 2006 Feb 7;47(3):605-10. doi: 10.1016/j.jacc.2005.09.035. Epub 2006 Jan 18. PMID 16458144
- [Background] Jung PH, Rieber J, Stork S, Hoyer C, Erhardt I, Nowotny A, Voelker W, Weidemann F, Ertl G, Klauss V, Angermann CE. Effect of contrast application on interpretability and diagnostic value of dobutamine stress echocardiography in patients with intermediate coronary lesions: comparison with myocardial fractional flow reserve. Eur Heart J. 2008 Oct;29(20):2536-43. doi: 10.1093/eurheartj/ehn204. Epub 2008 May 21. PMID 18499651
- [Background] Weidemann F, Jung P, Hoyer C, Broscheit J, Voelker W, Ertl G, Stork S, Angermann CE, Strotmann JM. Assessment of the contractile reserve in patients with intermediate coronary lesions: a strain rate imaging study validated by invasive myocardial fractional flow reserve. Eur Heart J. 2007 Jun;28(12):1425-32. doi: 10.1093/eurheartj/ehm082. Epub 2007 May 15. PMID 17504804
- [Background] Samady H, Lepper W, Powers ER, Wei K, Ragosta M, Bishop GG, Sarembock IJ, Gimple L, Watson DD, Beller GA, Barringhaus KG. Fractional flow reserve of infarct-related arteries identifies reversible defects on noninvasive myocardial perfusion imaging early after myocardial infarction. J Am Coll Cardiol. 2006 Jun 6;47(11):2187-93. doi: 10.1016/j.jacc.2006.01.065. PMID 16750683
- [Background] Lachance P, Dery JP, Rodes-Cabau J, Potvin JM, Barbeau G, Bertrand OF, Gleeton O, Larose E, Nguyen CM, Noel B, Proulx G, Roy L, De Larochelliere R. Impact of fractional flow reserve measurement on the clinical management of patients with coronary artery disease evaluated with noninvasive stress tests prior to cardiac catheterization. Cardiovasc Revasc Med. 2008 Oct-Dec;9(4):229-34. doi: 10.1016/j.carrev.2008.02.002. PMID 18928947
- [Background] Steinberg EH, Madmon L, Patel CP, Sedlis SP, Kronzon I, Cohen JL. Long-term prognostic significance of dobutamine echocardiography in patients with suspected coronary artery disease: results of a 5-year follow-up study. J Am Coll Cardiol. 1997 Apr;29(5):969-73. doi: 10.1016/s0735-1097(97)00032-6. PMID 9120183
- [Background] Danad I, Szymonifka J, Twisk JWR, Norgaard BL, Zarins CK, Knaapen P, Min JK. Diagnostic performance of cardiac imaging methods to diagnose ischaemia-causing coronary artery disease when directly compared with fractional flow reserve as a reference standard: a meta-analysis. Eur Heart J. 2017 Apr 1;38(13):991-998. doi: 10.1093/eurheartj/ehw095. PMID 27141095
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Pingitore A, Picano E, Varga A, Gigli G, Cortigiani L, Previtali M, Minardi G, Colosso MQ, Lowenstein J, Mathias W Jr, Landi P. Prognostic value of pharmacological stress echocardiography in patients with known or suspected coronary artery disease: a prospective, large-scale, multicenter, head-to-head comparison between dipyridamole and dobutamine test. Echo-Persantine International Cooperative (EPIC) and Echo-Dobutamine International Cooperative (EDIC) Study Groups. J Am Coll Cardiol. 1999 Nov 15;34(6):1769-77. doi: 10.1016/s0735-1097(99)00423-4. PMID 10577568
- [Background] Thomas D, Xie F, Smith LM, O'Leary E, Smith K, Olson J, Nalty K, Hess R, Graham M, Therrien S, Porter TR. Prospective randomized comparison of conventional stress echocardiography and real-time perfusion stress echocardiography in detecting significant coronary artery disease. J Am Soc Echocardiogr. 2012 Nov;25(11):1207-14. doi: 10.1016/j.echo.2012.08.016. Epub 2012 Sep 19. PMID 22998856